CLINICAL TRIAL: NCT05921045
Title: Shoulder Dystocia Delivery and Learning Skills on Mannequin
Brief Title: Learning Skills in Shoulder Dystocia Delivery Using Simulator Models
Status: Completed | Type: Observational
Sponsor: G. d'Annunzio University (Other)
Collaborators: Humanitas Hospital, Italy (Other); Federico Prefumo, Istituto Giannina Gaslini (Unknown); Claudio Meloni, University of Florence (Unknown)
Responsible Party: Principal Investigator, Claudio Celentano, Principal investigator, G. d'Annunzio University
Other Study IDs: ObGynEASC002
Record Dates: First submitted 2023-06-08; First posted 2023-06-27 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2023-07

CONDITIONS: Shoulder Dystocia - Delivered; Birth Disorder
Keywords: emergency delivery; Shoulder dystocia; mannequin
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Shoulder Dystocia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- time 0 and 6 months answers: questionnaire answers after first training and after re-training on shoulder dystocia model
  Interventions: Other: modification of clinical approach in clinical practice at time 0; Other: modification of clinical approach in clinical practice at 6 months

INTERVENTIONS:
Other: modification of clinical approach in clinical practice at time 0 — evaluation of modification in clinical approach after training
  Other Names: questionnaire for evaluation of modification in clinical approach
Other: modification of clinical approach in clinical practice at 6 months — evaluation of modification in clinical approach after retraining
  Other Names: questionnaire for evaluation of modification in clinical approach

SUMMARY:
Learning skills on shoulder dystocia on doctor and midwife

DETAILED DESCRIPTION:
Active learning on mannequin for shoulder dystocia deliveries on doctor and midwife using role play approach and its effect on clinical practice using questionnaires after first training and 6 months training

ELIGIBILITY:
Inclusion Criteria:

* residents and specialists in obstetrics and gynecology
* midwives

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: residents specialists midwies
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Management of SD | 6 months
  incidence of personal management of SD and fetal and neonatal outcomes in previous experiences and in successive

SECONDARY OUTCOMES:
Clinical approach in labor ward in identification and management of SD (with previous SD) | 6 months
  modification in approach if previous experience occurred
Clinical approach in labor ward in identification and management of SD (without previous SD) | 6 months
  modification in approach without previous experience

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Celentano, MD, Principal Investigator — EASC
Locations (1):
- Claudio Celentano, Pescara, Italia, Italy

IPD SHARING:
Plan to Share IPD: Undecided
recruiting residents, specialists and midwives in University of Chieti and Pescara Hospital